CLINICAL TRIAL: NCT05225688
Title: Skeletal Muscle Structure and Function in Relation to Post-exertional Malaise in Patients With PASC and ME/CFS
Brief Title: Skeletal Muscle in PASC and ME/CFS Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Patient-Led Research Collaborative Long COVID (Unknown)
Responsible Party: Principal Investigator, Michele van Vugt, Prof., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL78394.018.21
Record Dates: First submitted 2022-01-24; First posted 2022-02-04 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: LONG-COVID; Post-acute Sequelae of COVID-19; ME/CFS
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue Syndrome, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Frozen tissue, whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PASC patients: Non-hospitalized covid-19 patients with Post-acute Sequelae of COVID-19
  Interventions: Behavioral: Bike exertion test
- Healthy controls: Non-hospitalized covid-19 patients without residual symptoms
  Interventions: Behavioral: Bike exertion test
- ME/CFS patients: Patients with ME/CFS
  Interventions: Behavioral: Bike exertion test

INTERVENTIONS:
Behavioral: Bike exertion test — maximal exercise test

SUMMARY:
Rationale: A common feature in patients with Post-Acute Sequelae of SARS-CoV-2 Infection (PASC) and Myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS) are skeletal muscle-related symptoms, such as muscle pain, weakness, fatigue and post-exertional malaise.

Objective: The primary aim is to determine markers for skeletal muscle structure and function, and circulating factors, in patients with PASC and ME/CFS, and compare with controls. The secondary objective is to determine skeletal muscle structure and function before and after induction of post-exertional malaise, and assess the relationships between the measures obtained from muscle biopsies and parameters of exercise tolerance.

Study design: Case-control observational study

Study population: Patients with PASC, ME/CFS and healthy human volunteers, 18 - 65 yr old.

Intervention (if applicable): none

Main study parameters/endpoints: Primary outcome parameters are markers for local inflammation, viral infiltration, mitochondrial respiratory function and myokine concentrations in a muscle biopsy and venous blood before and after induction of post-exertional malaise. Heart rate variability and measures of exercise performance will also be determined.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participants will be asked to perform physical exercise tests, give muscle biopsies (2 samples), and various blood samples. There is some extent of burden and risk associated with harvesting muscle biopsies and blood samples, however this will be mitigated by the fact that these procedures will only be carried out by trained physicians. Moreover, the scientific gain from obtaining intracellular information outweighs these relatively quick procedures with minimal discomfort afterwards. The acute risks of the physical exercise measurements are negligible. The main risk for patients is that these patients often suffer from post-exertional malaise, which causes the participants to feel fatigued for some time after the maximal exercise test. It is one of the aims to better understand post-exertional malaise.

DETAILED DESCRIPTION:
1. INTRODUCTION AND RATIONALE Post-Acute Sequelae of SARS-CoV-2 Infection (PASC) and Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS) are severely debilitating diseases mainly characterized by chronic fatigue, post-exertional malaise (PEM) and cognitive impairment with autonomic, neuro-endocrine, immunological and cognitive involvement(Davis et al. 2021; Deumer et al. 2021; Soares et al. 2022). The clinical presentation of both diseases is remarkably overlapping. Particularly, skeletal muscle-related complaints, such as extreme fatigue, muscle weakness and muscle pain, are symptoms that tremendously decrease the patients quality of life and overlap in both patient groups, The key symptom, PEM, distinguishes PASC and ME/CFS from other more common fatigue conditions and is characterized by worsening or relapse of symptoms (including sleep dysfunction, cognitive impairment and extreme skeletal muscle fatigue) after physical activity, which can last for days or weeks(Davis et al. 2021; Soares et al. 2022; Stussman et al. 2020). We recently reviewed the skeletal muscle alterations in both acute SARS-CoV-2 infection and patients with Long COVID, and concluded that post-exertional malaise in patients with Long COVID cannot be explained by current knowledge on skeletal muscle structure and function(Soares et al. 2022).

   A possible lead to the understanding of PEM in Long COVID and ME/CFS pathophysiology is provided by the observation that most cases appear to have an infectious onset(Choutka et al. 2022; Magnus et al. 2015; Tsai et al. 2014). Following SARS-CoV-2 infection, 10-30% of patients exhibit post-infectious fatigue syndrome, called Long COVID or post-COVID condition(Ballering et al. 2022). PEM is the hallmark symptom of Long COVID and ME/CFS and a criterion for CCC, ICCC and IOM case definitions. Little is known about the underlying pathophysiology of skeletal muscle abnormalities, including PEM. No treatment options are available, apart from the advice to patients to avoid exercise or exercise below an (unknown) threshold.

   Due to the heterogeneity of patients, these muscle-related symptoms may vary dramatically, and is likely multifactorial in nature. Whilst long-term consequences of hospitalization are known, the widespread incidence of muscle-related symptoms suggests that skeletal muscle adaptations seen in non-hospitalized patients with PASC and ME/CFS stand apart from those seen in critical illness myopathy.

   The muscle weakness can range from mild to severe, and such symptoms may persist long after the viral infection has resolved. The high prevalence of skeletal muscle-related symptoms hint towards structural and functional alterations in skeletal muscle in patients with PASC and ME/CFS(Kerkhoff et al. 2022; McGregor et al. 2019; Noor et al. 2021). In this study, we aim to study alterations in intracellular skeletal muscle structure and function and the immune response that will help to explain why patients with PASC and ME/CFS suffer from post-exertional fatigue.
2. OBJECTIVES

   To obtain insight whether skeletal muscle adaptations can explain post-exertional fatigue malaise in patients with PASC and ME/CFS, the present study will address the following objectives:

   Primary objectives:

   • To determine markers for skeletal muscle structure and function (such as mitochondrial ultrastructure and function, viral infiltration, metabolite concentrations, myokine secretion), the immune response and circulating myokines (muscle-derived molecules), in non-hospitalized patients with PASC, ME/CFS and healthy controls.

   Secondary objectives:

   • To determine each of the above variables both before and after induction of post-exertional malaise, and assess the relationships between the measures obtained from muscle biopsies and parameters of exercise tolerance.
3. STUDY DESIGN 3.1. General. Case-control study with assessments before and after an induction of post-exertional malaise. 26 PASC patients, 26 ME/CFS patients and 30 matched healthy controls who have recovered from a SARS-COV-2 infection will be recruited for the study. Participants are required to visit the laboratory for a total of 5 experimental sessions, for a total duration of approximately 8 hours. Four measurements will take place within a time window of 2 weeks. On day 10, patients will fill in a digital questionnaire. The last time point will be 1 year after the start of the study. See Figure 1 for an overview of study design.

26 participants with PASC and 26 patients with ME/CFS (equal split between sexes) between the ages of 18-65 yrs will be recruited for the study. 30 healthy participants matched for age BMI and preferably physical activity levels will be included as a control group

Participants will be required to visit the laboratory on 4 separate occasions over a 2 week period immediately prior to and following a maximal exercise test. One year (± three months) we will require one additional visit. After the first visit, participants will be asked to confirm dates for the subsequent visits over the next 2 weeks face-to-face in the laboratory. Participants will be instructed not to consume alcohol or perform strenuous exercise within the 24 h preceding each exercise test, and to abstain from caffeine consumption for at least 3 h.

4. STUDY POPULATION

4.1 Population 26 non-hospitalized participants with diagnosed PASC, 26 ME/CFS patients and 30 healthy participants of similar sex, age, BMI and preferably current physical activity levels between the ages of 18-65 years old will be recruited to the study. All participants with PASC will be recruited from the outpatient clinic of the Amsterdam UMC, ME/CFS patients will be recruited through ME/CFS specialists in the Netherlands, whereas healthy controls will be recruited via specific social media groups, through personal networks and/or posters. All testing will be conducted at the Faculty of Behavioural and Movement Sciences, Vrije Universiteit Amsterdam, Amsterdam under the direct supervision of BA or MvV from the Amsterdam UMC. Therefore, participants should be currently residing in or willing to travel to Amsterdam.

ELIGIBILITY:
Inclusion criteria

In order to be eligible to participate in this study, a subject with PASC must meet all of the following criteria:

* Non-hospitalized individuals with prior confirmed diagnosis of severe acute respiratory coronavirus 2 (SARS-CoV-2) infection by reverse transcription-polymerase chain reaction testing or serology (wantai) testing
* Individuals with diagnosed PASC by a post-covid physician
* >3 months of symptoms
* Post exertional malaise, according to the DSQ-PEM questionnaire or 1:1 interview with post-covid physician
* No symptoms present before confirmed diagnosis of severe acute respiratory coronavirus 2
* Aged between 18-65 years

In order to be eligible to participate in this study, a subject with ME/CFS must meet all of the following criteria:

* Fulfill the Canadian Consensus Criteria (CCC)
* Post exertional malaise, according to the DSQ-PEM questionnaire or 1:1 interview with post-covid physician
* >3 months of symptoms
* Aged between 18-65 years
* Confirmed diagnosis of severe acute respiratory coronavirus2 (SARS-CoV-2) infection by reverse transcription-polymerase chain reaction testing or serology (wantai) testing

For the healthy controls:

* Aged between 18-65 years
* Confirmed diagnosis of severe acute respiratory coronavirus2 (SARS-CoV-2) infection by reverse transcription-polymerase chain reaction testing or serology (wantai) testing without admission

Exclusion criteria

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* History of asthma, stroke, chronic obstructive pulmonary disease, congestive heart failure, heart surgery, or congenital heart diseases
* Severe illness (e.g., active malignancy, CHD, uncontrolled diabetes)
* Current treatment with drugs known to interfere with metabolism e.g. systemic corticosteroids, statins, SGLT2 inhibitors, GLP1 receptor agonists or immune modulatory drugs in the last three months.
* Severe psychiatric or mood disorders
* Insulin pump therapy
* Symptomatic autonomic or distal neuropathy
* BMI >35 due to adiposity, since this is known to cause difficulties in obtaining muscle biopsies.
* Pregnancy
* Recent acute myocardial infarction (<6 months)
* Uncontrolled arrhythmia/severe conduction disorder (atrial fibrillation or second/third degree AV block) causing hemodynamic compromise
* Implantable pacemaker or other cardiac device with complete ventricular pacing
* Uncontrolled heart failure with hemodynamic compromise
* Uncontrolled hypertension (Systolic Blood Pressure >150 mmHg and Diastolic Blood Pressure > 100 mmHg on repeated measurements)
* Active infection, anaemia, severe renal dysfunction (estimated Glomerular filtration rate <30 ml/min/1,73m2) likely to significantly impact on exercise performance
* Chronic illness (including orthopaedic, endocrinological, haematological, malignant, gastrointestinal, neurological, muscle or inflammatory disorders) likely to significantly impact on exercise performance
* > 6 alcohol units per day or >14 alcohol units per week
* Use of anticoagulants or anti platelet therapy

For the healthy controls:

● Individuals hospitalized in the last 6 months (i.e. after SARS-CoV-2 infection).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 26 non-hospitalized participants with diagnosed PASC, 26 patients with ME/CFS and 30 healthy participants of similar sex, age, BMI and preferably current physical activity levels between the ages of 18-65 years old will be recruited to the study.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Skeletal muscle mitochondrial respiratory function | 7 days
Local and systemic inflammation markers after induction of post-exertional malaise | 14 days

SECONDARY OUTCOMES:
Heart rate variability during post-exertional malaise in LONG-COVID patients | 14 days
Exercise tolerance in LONG-COVID patients. | 7 days
Muscle oxygenation derived via near-infrared spectroscopy (NIRS) during exercise in LONG-COVID patients | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam university medical centre AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Appelman B, Charlton BT, Goulding RP, Kerkhoff TJ, Breedveld EA, Noort W, Offringa C, Bloemers FW, van Weeghel M, Schomakers BV, Coelho P, Posthuma JJ, Aronica E, Joost Wiersinga W, van Vugt M, Wust RCI. Muscle abnormalities worsen after post-exertional malaise in long COVID. Nat Commun. 2024 Jan 4;15(1):17. doi: 10.1038/s41467-023-44432-3. PMID 38177128